CLINICAL TRIAL: NCT00883753
Title: An Extension Phase of the Multi-National Open-Label Study (MA21573) to Evaluate the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs Who Have an Inadequate Response to Current Non-biologic DMARD and/or Anti-TNF Therapy.
Brief Title: An Extension to Study MA21573, Evaluating Tocilizumab in Patients With Active Rheumatoid Arthritis and an Inadequate Response to Current Non-Biological DMARDs and/or Anti-tumor Necrosis Factor (TNF) Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA22460; 2008-006924-68
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- tocilizumab (Experimental): Participants received tocilizumab 8 mg/kg intravenous (IV), maximum dose not exceeding 800 mg in a single infusion, every 4 weeks for up to 104 weeks or up to 4 weeks after tocilizumab became commercially available in the respective country whichever occurred first.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg IV (maximum dose not exceeding 800 mg in a single infusion) every 4 weeks.

SUMMARY:
This study was an extension to study MA21573 [NCT00750880], which was an open label single arm study to investigate the safety, tolerability and efficacy of tocilizumab monotherapy, or combination therapy with non-biological disease-modifying antirheumatic drugs (DMARDS), in patients with moderate to severe active rheumatoid arthritis. Patients who completed the 24 week core study, and had at least a moderate European League Against Rheumatism (EULAR) response, were eligible to enter this long-term extension study, and received tocilizumab 8 mg/kg intravenous (iv) every 4 weeks. The anticipated time on study treatment was 1-2 years, and the target sample size was > 500 individuals.

ELIGIBILITY:
Inclusion Criteria:

- patients who completed the 24-week MA21573 core study, had at least a moderate response based on EULAR definition criteria and no adverse events (AEs), serious adverse events (SAEs) or conditions that led to unacceptable risk of continued treatment.

Exclusion Criteria:

-as for MA21573.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (152):
- Australia (8):
  - Canberra, Australian Capital Territory
  - Coffs Harbour, New South Wales
  - Kogarah, New South Wales
  - Cairns, Queensland
  - Adelaide, South Australia
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
- Canada (19):
  - Edmonton, Alberta
  - Lethbridge, Alberta
  - Kelowna, British Columbia
  - Nanaimo, British Columbia
  - Vancouver, British Columbia
  - Quispamsis, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Rimouski, Quebec
  - Saint-Eustache, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
- Czechia (6):
  - Bruntál
  - Ostrava
  - Prague
  - Sokolov
  - Uherské Hradiště
  - Zlín
- France (22):
  - Belfort
  - Caen
  - Cahors
  - Corbeil-Essonnes
  - Dijon
  - La Rochelle
  - Liévin
  - Lomme
  - Lyon
  - Marseille
  - Montivilliers
  - Montpellier
  - Mulhouse
  - Paris
  - Poitiers
  - Reims
  - Roubaix
  - Saint-Brieuc
  - Strasbourg
  - Toulouse
  - Valence
  - Valenciennes
- Heraklion, Greece
- Hungary (4):
  - Budapest
  - Eger
  - Szeged
  - Veszprém
- Italy (11):
  - Arenzano
  - Legnano
  - Milan
  - Modena
  - Monserrato
  - Novara
  - Palermo
  - Potenza
  - Roma
  - Siena
  - Varese
- Netherlands (20):
  - 's-Hertogenbosch
  - Alkmaar
  - Amsterdam
  - Apeldoorn
  - Arnhem
  - Bergen op Zoom
  - Den Helder
  - Enschede
  - Flushing
  - Gouda
  - Heerlen
  - Hilversum
  - Leeuwarden
  - Nieuwegein
  - Nijmegen
  - Roosendaal
  - Rotterdam
  - Schiedam
  - Spijkenisse
  - The Hague
- Poland (3):
  - Krakow
  - Poznan
  - Wroclaw
- Portugal (4):
  - Almada
  - Coimbra
  - Lisbon
  - Porto
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Jeddah, Saudi Arabia
- Spain (20):
  - Alicante, Alicante
  - Elche, Alicante
  - Elda, Alicante
  - Almería, Almeria
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Cáceres, Caceres
  - Córdoba, Cordoba
  - Granada, Granada
  - Huesca, Huesca
  - A Coruña, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - Lugo, Lugo
  - Madrid, Madrid
  - Málaga, Malaga
  - Salamanca, Salamanca
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia
- United Kingdom (31):
  - Barnsley
  - Basingstoke
  - Bournemouth
  - Brighton
  - Burton-on-Trent
  - Bury Saint Edmonds
  - Cambridge
  - Cardiff
  - Chelmsford
  - Dudley
  - Eastbourne
  - Gillingham
  - Harrogate
  - Ipswich
  - Liverpool
  - Llantrisant
  - London
  - Londonderry
  - Maidstone
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - Newcastle upon Tyne
  - Nottingham
  - Reading
  - Salford
  - Sheffield
  - Southport
  - Swindon
  - Torquay
  - Westcliffe-on-sea
  - Worthing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients participated in the 24 Week Core Study: MA21573 [NCT00750880] then continued to receive tocilizumab in this extension study for total treatment time of up to 104 weeks + a 4 week follow-up.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 934
Completed | 827
Not Completed | 107
Not completed — Adverse Event | 37
Not completed — Death | 2
Not completed — Insufficient therapeutic response | 16
Not completed — Lost to Follow-up | 4
Not completed — Violation of selection criteria at entry | 7
Not completed — Protocol Violation | 2
Not completed — Refused treatment | 4
Not completed — Withdrew consent | 10
Not completed — Investigator's decision | 17
Not completed — Administrative/Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 753
  Male | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant. The percentage of participants with AEs and SAEs that occurred in the Extension Study grouped according to the number of disease-modifying anti-rheumatic drugs (DMARD) a participant was taking at Core Baseline is presented.
Time Frame: 108 Weeks
Population: LTE Safety population included all participants who received study drug and had at least one assessment of safety in the long term extension (LTE).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tocilizumab Monotherapy: Participants received tocilizumab 8 mg/kg IV, maximum dose not exceeding 800 mg in a single infusion, every 4 weeks for up to 104 weeks or up to 4 weeks after tocilizumab became commercially available in the respective country whichever occurred first, in a subset of patients who were not taking DMARDS at Core Baseline.
- Tocilizumab + 1 DMARD: Participants received tocilizumab 8 mg/kg IV, maximum dose not exceeding 800 mg in a single infusion, every 4 weeks for up to 104 weeks or up to 4 weeks after tocilizumab became commercially available in the respective country whichever occurred first, in a subset of patients who were taking one DMARD at Core study Baseline.
- Tocilizumab + > 1 DMARD: Participants received tocilizumab 8 mg/kg IV, maximum dose not exceeding 800 mg in a single infusion, every 4 weeks for up to 104 weeks or up to 4 weeks after tocilizumab became commercially available in the respective country whichever occurred first, in a subset of patients who were taking more than one DMARD at Core study Baseline.
Arm/Group | Tocilizumab Monotherapy | Tocilizumab + 1 DMARD | Tocilizumab + > 1 DMARD
Number analyzed (Participants) | 117 | 612 | 205
percentage of participants
  AEs | 65.0 [55.6 to 73.5] | 68.6 [64.8 to 72.3] | 73.2 [66.6 to 79.1]
  SAEs | 8.5 [4.2 to 15.2] | 5.7 [4.0 to 7.9] | 7.3 [4.2 to 11.8]

2. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Withdraw
Description: An Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV, maximum dose not exceeding 800 mg in a single infusion, every 4 weeks for up to 104 weeks or up to 4 weeks after tocilizumab became commercially available in the respective country whichever occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants | 4.0 [2.7 to 5.3]

3. Secondary Outcome: Time to Withdrawal Due to an Adverse Event (AE)
Description: Time to withdrawal was defined as the number of days from Core Study Day 1 to the first date of onset of the AE leading to discontinuation of tocilizumab.
Time Frame: 108 Weeks
Population: LTE Safety population included all participants who received study drug and had at least one assessment of safety in the long term extension(LTE). Participants who did not experience an AE-related treatment discontinuation of tocilizumab were censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
days | 374.5 [286.0 to 441.0]

4. Secondary Outcome: Percentage of Participants With Discontinuation of Treatment Due to Any Cause
Description: Percentage of participants who discontinued treatment with tocilizumab for any reason.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants | 11.5

5. Secondary Outcome: Time to Discontinuation of Tocilizumab Treatment for Any Cause
Description: Time in days from start of the Core Study Day 1 to discontinuation of tocilizumab for any reason.
Time Frame: 108 Weeks
Population: LTE Safety population included all participants who received study drug and had at least one assessment of safety in the long term extension (LTE). Participants who did not experience discontinuation of tocilizumab treatment were censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
days | 339.0 [294.0 to 370.0]

6. Secondary Outcome: Percentage of Participants With Marked Lipid Abnormalities
Description: Fasting blood samples were collected for Lipids: Cholesterol, Triglyceride, High-density lipoprotein (HDL) Cholesterol, Low-density lipoprotein (LDL) Cholesterol every 12 weeks and at follow-up in the Extension study and were sent to a central laboratory for analysis. Lipid abnormalities were defined as a High Cholesterol, High Triglyceride, Low HDL Cholesterol and a High LDL Cholesterol that occurred at any time in the extension study.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Cholesterol (high) | 4.2
  HDL Cholesterol (low) | 0.0
  LDL Cholesterol (high) | 6.5
  Triglyceride (high) | 14.9

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) of Special Interest
Description: An Adverse Event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events. Adverse Events of special interest for this study were: Infections (preferred term in the infection adverse event group term), Serious Infections (an infection that qualified as Serious Adverse Event), Infusion Reactions (occurred during infusion or within 24 hours of infusion), Major Cardiac AE (Myocardial Infarction/ Acute Coronary Syndrome), Stroke or Death.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Infections | 40.4
  Serious Infections | 2.4
  Infusion Reaction | 2.9
  Major Cardiac AE | 0.3
  Stroke | 0.9
  Death | 0.3

8. Secondary Outcome: Percentage of Participants With ALT Elevations > 3*ULN
Description: Blood samples were collected for the Liver Function Test: Alanine aminotransferase (ALT) every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. Percentage of participants with any values greater than 3 times the Upper Limit of Normal (3*ULN) is reported. ULN= 55 Units/Liter.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants | 1.9

9. Secondary Outcome: Percentage of Participants With AST Elevations > 3*ULN
Description: Blood was collected for the Liver Function Test: Aspartate aminotransferase (AST) every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. Percentage of participants with any values greater than 3 times the Upper Limit of Normal (3*ULN) is reported. ULN= 40 Units/Liter.
Time Frame: 108 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants | 0.4

10. Secondary Outcome: Number of Participants Categorized by Highest Value for ALT (SGPT) During the Study
Description: Blood samples were collected for liver function test: Alanine aminotransferase (serum glutamic-pyruvic transaminase) [ALT(SGPT)] every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. The Upper Limit of Normal (ULN) for ALT=55 Units/Liter. The number of participants categorized by the highest value for ALT/GPT during the study is reported: Normal (ALT result within the central lab reference range), Greater than the ULN to 1.5 times the ULN (>ULN to 1.5*ULN), 1.5 times the ULN to 3 times the ULN (1.5*ULN to 3*ULN) and 3 times the ULN to 5 times the ULN (3*ULN to 5*ULN).
Time Frame: 108 Weeks
Population: Participants from the LTE Safety population included all participants who received study drug and had at least one assessment of safety in the long term extension (LTE) with data available for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
participants
  Normal | 874
  >ULN - 1.5*ULN | 50
  1.5*ULN to 3*ULN | 8
  3*ULN to 5*ULN | 2

11. Secondary Outcome: Number of Participants Categorized by Worst Value for AST (SGOT) During the Study
Description: Blood samples were collected for liver function test: Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase) [AST (SGOT)] every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. The Upper Limit of Normal (ULN) for AST=40 Units/Liter. The number of participants categorized by worst value for AST(SGOT) during the study is reported: Normal (AST result is within the central lab reference range), Greater than the ULN to 1.5 times the ULN (>ULN to 1.5*ULN), 1.5 times the ULN to 3 times the ULN (1.5*ULN to 3*ULN) and 3 times the ULN to 5 times the ULN (3*ULN to 5*ULN).
Time Frame: 108 Weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
participants
  Normal | 903
  >ULN to 1.5*ULN | 26
  1.5*ULN to 3*ULN | 4
  3*ULN to 5*ULN | 1

12. Secondary Outcome: Number of Participants Categorized by Worst Value for LDL Cholesterol During the Study
Description: Blood samples were collected for LDL Cholesterol every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. The number of participants categorized by the worst value for LDL Cholesterol during the study is reported: Low is below central lab reference range, Normal is within the central lab reference range and High is above central lab reference range.
Time Frame: 108 Weeks
Population: Participants from the LTE Safety population (all participants who received study drug and had at least one assessment of safety in the long term extension) with data available for analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 933
participants
  Low | 0
  Normal | 368
  High | 565

13. Secondary Outcome: Number of Participants Categorized by Worst Value for Total Cholesterol During the Study
Description: Blood samples were collected for Total Cholesterol every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. The number of participants categorized by worst value for Total Cholesterol during the study is reported: Low is below central lab reference range, Normal is within the central lab reference range and High is above central lab reference range.
Time Frame: 108 Weeks
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 933
participants
  Low | 4
  Normal | 194
  High | 735

14. Secondary Outcome: Number of Participants Categorized by Worst Value for Neutrophil Count During the Study
Description: Blood samples were collected for a Neutrophil Count every 12 weeks and at the follow-up visit in the Extension study and were sent to a central laboratory for analysis. The number of participants categorized by the worst value for Neutrophil Count during the study is reported: Low is below central lab reference range, Normal is within the central lab reference range and High is above central lab reference range.
Time Frame: 108 Weeks
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 932
participants
  Low | 321
  Normal | 608
  High | 3

15. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement in Disease Activity Score-28 (DAS28)
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. Clinical meaningful improvement was defined as a ≥ 1.2 unit reduction in DAS28.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: Long Term Extension Intent-to-treat (LTE ITT) population included all participants from the Core Study who received at least one dose of study drug in the Extension Study. "n" in each of the categories is the number of participants with data available for both Baseline and the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 (n=889) | 94.7
  Week 24 (n=757) | 94.8
  Week 36 (n=607) | 96.4
  Week 48 (n=440) | 96.6
  Week 60 (n=320) | 97.8
  Week 72 (n=216) | 96.8
  Week 84 (n=119) | 95.8
  Week 96 (n=54) | 100.0
  Week 108 (n=42) | 100.0

16. Secondary Outcome: Percentage of Participants With DAS28 Low Disease Activity
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. Low Disease Activity was defined as a score of < 3.2.
Time Frame: Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: LTE ITT population included all participants from the Core Study who received at least one dose of study drug in the Extension Study. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 (n=891) | 75.3
  Week 24 (n=759) | 76.9
  Week 36 (n=609) | 77.3
  Week 48 (n=440) | 78.2
  Week 60 (n=320) | 80.6
  Week 72 (n=216) | 84.3
  Week 84 (n=119) | 83.2
  Week 96 (n=54) | 88.9
  Week 108 (n=42) | 83.3

17. Secondary Outcome: Percentage of Participants With DAS28 Remission
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission was defined as a DAS28 score < 2.6.
Time Frame: Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 (n=891) | 59.6
  Week 24 (n=759) | 61.9
  Week 36 (n=609) | 62.7
  Week 48 (n=440) | 62.7
  Week 60 (n=320) | 65.9
  Week 72 (n=216) | 69.9
  Week 84 (n=119) | 68.9
  Week 96 (n=54) | 70.4
  Week 108 (n=42) | 71.4

18. Secondary Outcome: Change From Baseline in DAS28
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: LTE ITT population included all participants from the Core Study who received at least one dose of study drug in the Extension Study. "n" in each of the categories is the number of participants with data available at both Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=889) | -3.58 (1.498)
  Week 24 (n=757) | -3.62 (1.496)
  Week 36 (n=607) | -3.74 (1.443)
  Week 48 (n=440) | -3.80 (1.420)
  Week 60 (n=320) | -3.91 (1.318)
  Week 72 (n=216) | -3.93 (1.394)
  Week 84 (n=119) | -3.94 (1.273)
  Week 96 (n=54) | -4.14 (1.132)
  Week 108 (n=42) | -4.12 (1.178)

19. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: 68 joints were assessed for tenderness and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
joint count
  Week 12 (n=927) | -17.45 (14.492)
  Week 24 (n=789) | -18.07 (14.524)
  Week 36 (n=627) | -18.592 (14.59)
  Week 48 (n=457) | -18.77 (14.744)
  Week 60 (n=334) | -19.16 (13.575)
  Week 72 (n=223) | -18.30 (13.157)
  Week 84 (n=121) | -17.45 (12.481)
  Week 96 (n=55) | -17.47 (11.445)
  Week 108 (n=43) | -17.35 (12.049)

20. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: 66 joints were assessed for swelling and joints were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
joint count
  Week 12 (n=927) | -10.16 (9.838)
  Week 24 (n=789) | -10.17 (9.633)
  Week 36 (n=627) | -10.55 (9.981)
  Week 48 (n=457) | -10.78 (10.410)
  Week 60 (n=334) | -10.83 (8.885)
  Week 72 (n=223) | -10.91 (8.563)
  Week 84 (n=121) | -9.90 (6.378)
  Week 96 (n=55) | -8.62 (7.230)
  Week 108 (n=43) | -8.58 (5.662)

21. Secondary Outcome: Change From Baseline in Patient Assessment of Pain Visual Analog Scale (VAS)
Description: The patient assessed their pain using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
mm
  Week 12 (n=900) | -32.52 (26.297)
  Week 24 (n=772) | -32.59 (25.998)
  Week 36 (n=612) | -33.04 (25.461)
  Week 48 (n=445) | -32.69 (27.244)
  Week 60 (n=326) | -35.35 (26.082)
  Week 72 (n=219) | -35.24 (27.901)
  Week 84 (n=119) | -35.71 (25.901)
  Week 96 (n=55) | -43.40 (21.131)
  Week 108 (n=42) | -45.48 (20.956)

22. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity VAS
Description: The patients global assessment of disease activity was assessed on a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=900) | -35.90 (25.964)
  Week 24 (n=773) | -35.57 (25.368)
  Week 36 (n=612) | -35.75 (25.853)
  Week 48 (n=445) | -35.56 (27.475)
  Week 60 (n=326) | -37.85 (26.723)
  Week 72 (n=219) | -36.36 (26.828)
  Week 84 (n=119) | -37.91 (27.628)
  Week 96 (n=55) | -45.44 (21.766)
  Week 108 (n=42) | -44.90 (28.689)

23. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity VAS
Description: The physician global assessment of disease activity was assessed using a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
mm
  Week 12 (n=900) | -41.14 (21.221)
  Week 24 (n=769) | -40.86 (21.114)
  Week 36 (n=613) | -40.97 (21.244)
  Week 48 (n=447) | -42.20 (21.551)
  Week 60 (n=325) | -42.67 (21.656)
  Week 72 (n=217) | -43.74 (20.941)
  Week 84 (n=119) | -42.68 (21.307)
  Week 96 (n=55) | -43.60 (17.828)
  Week 108 (n=42) | -44.38 (25.580)

24. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR) (a test that assesses tissue inflammation) and was analyzed at a local laboratory. ESR was measured in millimeters/hour (mm/hr). A reduction in the level is considered an improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: LTE ITT population included all participants from the Core Study who received at least one dose of study drug in the Extension Study. "n" in each of the categories is the number of participants with data available at Baseline and the given time-point.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
mm/hr
  Week 12 (n=903) | -30.59 (24.839)
  Week 24 (n=764) | -29.96 (24.584)
  Week 36 (n=615) | -31.56 (24.293)
  Week 48 (n=443) | -31.09 (24.408)
  Week 60 (n=320) | -31.61 (22.864)
  Week 72 (n=217) | -29.62 (21.904)
  Week 84 (n=119) | -29.79 (19.525)
  Week 96 (n=55) | -34.38 (18.865)
  Week 108 (n=42) | -36.67 (17.167)

25. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: Blood was collected for C-Reactive Protein (CRP) (a test for analysis of inflammatory and infectious disorders) and was analyzed at a central laboratory. The serum concentration of CRP was measured in milligrams/deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
mg/dL
  Week 12 (n=904) | -1.72 (2.785)
  Week 24 (n=767) | -1.73 (2.620)
  Week 36 (n=611) | -1.79 (2.756)
  Week 48 (n=445) | -1.73 (2.696)
  Week 60 (n=319) | -1.82 (2.823)
  Week 72 (n=208) | -1.54 (2.609)
  Week 84 (n=112) | -1.56 (2.618)
  Week 96 (n=54) | -1.24 (1.999)
  Week 108 (n=43) | -0.98 (1.324)

26. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR20) Response
Description: ACR20 response was defined as a ≥ 20 % improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 | 76.1
  Week 24 (n=827) | 75.1
  Week 36 (n=685) | 72.6
  Week 48 (n=534) | 69.1
  Week 60 (n=419) | 65.6
  Week 72 (n=313) | 60.7
  Week 84 (n=217) | 46.1
  Week 96 (n=154) | 31.8
  Week 108 (n=142) | 28.2

27. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50 (ACR50) Response
Description: ACR50 response is defined as a ≥ 50 % improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Core Baseline, Extension Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 | 56.3
  Week 24 (n=827) | 53.9
  Week 36 (n=685) | 53.6
  Week 48 (n=534) | 48.5
  Week 60 (n=419) | 49.2
  Week 72 (n=313) | 46.0
  Week 84 (n=217) | 33.2
  Week 96 (n=154) | 26.6
  Week 108 (n=142) | 23.9

28. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70 (ACR70) Response
Description: ACR70 response is defined as a ≥ 70 % improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 | 31.4
  Week 24 (n=827) | 31.0
  Week 36 (n=685) | 32.6
  Week 48 (n=534) | 31.3
  Week 60 (n=419) | 28.2
  Week 72 (n=313) | 29.7
  Week 84 (n=217) | 23.5
  Week 96 (n=154) | 20.8
  Week 108 (n=142) | 17.6

29. Secondary Outcome: Percentage of Participants With American College of Rheumatology 90 (ACR90) Response
Description: ACR90 response is defined as a ≥ 90 % improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 | 9.9
  Week 24 (n=827) | 10.5
  Week 36 (n=685) | 12.0
  Week 48 (n=534) | 11.2
  Week 60 (n=419) | 11.0
  Week 72 (n=313) | 11.2
  Week 84 (n=217) | 11.5
  Week 96 (n=154) | 9.7
  Week 108 (n=142) | 9.2

30. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Response
Description: The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A patient must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=895) | -0.58 (0.605)
  Week 24 (n=765) | -0.59 (0.611)
  Week 36 (n=611) | -0.61 (0.607)
  Week 48 (n=446) | -0.63 (0.595)
  Week 60 (n=327) | -0.65 (0.614)
  Week 72 (n=218) | -0.64 (0.610)
  Week 84 (n=119) | -0.68 (0.650)
  Week 96 (n=55) | -0.82 (0.582)
  Week 108 (n=42) | -0.87 (0.634)

31. Secondary Outcome: Percentage of Participants Achieving Clinical Meaningful Health Assessment Questionnaire Disability Index (HAQ-DI) Response
Description: The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A patient must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). Clinically meaningful improvement is defined as a reduction from Baseline in the HAQ-DI score ≥ 0.2.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 (n=895) | 73.6
  Week 24 (n=765) | 73.9
  Week 36 (n=611) | 74.1
  Week 48 (n=446) | 76.5
  Week 60 (n=327) | 76.8
  Week 72 (n=218) | 77.5
  Week 84 (n=119) | 76.5
  Week 96 (n=55) | 89.1
  Week 108 (n=42) | 90.5

32. Secondary Outcome: Percentage of Participants Achieving Health Assessment Questionnaire Disability Index (HAQ-DI) Clinical Remission
Description: The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A patient must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). Clinical Remission is defined as a HAQ-DI score < 0.5.
Time Frame: Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
percentage of participants
  Week 12 (n=900) | 32.1
  Week 24 (n=770) | 33.4
  Week 36 (n=614) | 34.5
  Week 48 (n=446) | 33.2
  Week 60 (n=327) | 37.0
  Week 72 (n=218) | 34.9
  Week 84 (n=119) | 38.7
  Week 96 (n=55) | 41.8
  Week 108 (n=42) | 50.0

33. Secondary Outcome: Change From Baseline in Quality of Life Short Form (SF-36): Physical Component Score
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=885) | 9.86 (10.548)
  Week 24 (n=747) | 9.30 (10.291)
  Week 36 (n=607) | 9.54 (10.580)
  Week 48 (n=444) | 9.82 (11.025)
  Week 60 (n=324) | 10.34 (10.837)
  Week 72 (n=217) | 10.38 (11.157)
  Week 84 (n=117) | 10.62 (10.378)
  Week 96 (n=55) | 13.06 (9.175)
  Week 108 (n=42) | 13.59 (9.932)

34. Secondary Outcome: Change From Baseline in Quality of Life Short Form (SF-36):Mental Component Score
Description: as for outcome 33
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: LTE ITT population included all participants from the Core Study who received at least one dose of study drug in the Extension Study. "n" in each of the categories is the number of participants with data available for both Baseline and at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=885) | 8.10 (14.426)
  Week 24 (n=747) | 8.37 (14.607)
  Week 36 (n=607) | 9.43 (14.311)
  Week 48 (n=444) | 8.27 (13.868)
  Week 60 (n=324) | 9.67 (13.91)
  Week 72 (n=217) | 8.30 (13.515)
  Week 84 (n=117) | 7.36 (14.466)
  Week 96 (n=55) | 10.57 (14.365)
  Week 108 (n=42) | 7.42 (12.272)

35. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status. A positive change from Baseline indicated improvement.
Time Frame: Core Baseline, Extension Weeks 12, 24, 36 ,48, 60, 72, 84, 96, 108
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 934
score on a scale
  Week 12 (n=900) | 10.67 (11.287)
  Week 24 (n=765) | 10.70 (11.239)
  Week 36 (n=613) | 11.42 (11.826)
  Week 48 (n=447) | 11.02 (11.684)
  Week 60 (n=326) | 11.77 (11.660)
  Week 72 (n=217) | 10.71 (11.170)
  Week 84 (n=119) | 10.63 (11.602)
  Week 96 (n=55) | 11.69 (10.374)
  Week 108 (n=42) | 10.56 (10.636)

ADVERSE EVENTS:
Time Frame: 108 Weeks
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 60/934
Other Adverse Events (participants affected / at risk) | 141/934
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=934)
Cellulitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 5
Diverticulitis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Cognitive Disorder (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient Ischaemic attack (Nervous system disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Device breakage (General disorders) | 1
Device dislocation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Thymus enlargement (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=934)
Nasopharyngitis (Infections and infestations) | 89
Upper respiratory tract infection (Infections and infestations) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.